CLINICAL TRIAL: NCT02024607
Title: A Phase Ib/II Clinical Study of BBI608 in Combination With Standard Chemotherapies in Adult Patients With Advanced Gastrointestinal Cancer
Brief Title: A Study of BBI608 in Combination With Standard Chemotherapies in Adult Patients With Advanced Gastrointestinal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBI608-246
Record Dates: First submitted 2013-12-20; First posted 2013-12-31 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Advanced Gastrointestinal Cancer
MeSH Terms: interventions — napabucasin; Fluorouracil; Oxaliplatin; Leucovorin; Irinotecan; Bevacizumab; Capecitabine; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- ARM A- BBI608 in combination with FOLFOX6 (Experimental): BBI608 is administered orally twice daily, continuously. Oxaliplatin 85 mg/m^2 together with leucovorin 400 mg/m^2 will be administered intravenously. 5-FU 400 mg/m^2 bolus will be administered intravenously immediately following oxaliplatin/leucovorin infusion, followed by 5-FU 1200 mg/m^2/day (total 2400 mg/m^2 over 46-48 hours) continuous intravenous infusion. This regimen will be repeated every 14 days thereafter.
  Interventions: Drug: BBI608; Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin
- ARM B- BBI608 in combination with FOLFOX6 and Bevacizumab (Experimental): BBI608 is administered orally twice daily, continuously. Oxaliplatin 85 mg/m^2 together with leucovorin 400 mg/m^2 will be administered intravenously. 5-FU 400 mg/m^2 bolus will be administered intravenously immediately following oxaliplatin/leucovorin infusion, followed by 5-FU 1200 mg/m^2/day (total 2400 mg/m^2 over 46-48 hours) continuous intravenous infusion. Bevacizumab 5 mg/kg will be administered intravenously following oxaliplatin/leucovorin infusion. This regimen will be repeated every 14 days thereafter.
  Interventions: Drug: BBI608; Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Bevacizumab
- ARM C- BBI608 in combination with CAPOX (Experimental): BBI608 is administered orally twice daily, continuously. CAPOX regimen will be administered orally (capecitabine) and IV (oxaliplatin). Capecitabine 850 mg/m^2 will be administered orally twice-daily for 14 consecutive days and be repeated every 21 days. Oxaliplatin will be administered IV and be repeated every 21 days thereafter. If capecitabine is tolerated at the 850 mg/m^2 twice daily dose, dosage may be increased to 1000 mg/m^2 twice daily as tolerated after the first cycle.
  Interventions: Drug: BBI608; Drug: Oxaliplatin; Drug: Capecitabine
- ARM D- BBI608 in combination with FOLFIRI (Experimental): BBI608 is administered orally twice daily, continuously. Irinotecan 180 mg/m^2 together with leucovorin 400 mg/m^2 will be administered intravenously. 5-FU 400 mg/m^2 bolus will be administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5-FU 1200 mg/m^2/day (total 2400 mg/m^2) continuous infusion. This regimen will be repeated every 14 days thereafter.
  Interventions: Drug: BBI608; Drug: Fluorouracil; Drug: Leucovorin; Drug: Irinotecan
- ARM E- BBI608 in combination with FOLFIRI and Bevacizumab (Experimental): BBI608 is administered orally twice daily, continuously. Irinotecan 180 mg/m^2 together with leucovorin 400 mg/m^2 will be administered intravenously 5-FU 400 mg/m^2 bolus will be administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5-FU 1200 mg/m^2/day (total 2400 mg/m^2) continuous infusion. Bevacizumab 5 mg/kg will be administered intravenously following oxaliplatin/leucovorin infusion. This regimen will be repeated every 14 days thereafter.
  Interventions: Drug: BBI608; Drug: Fluorouracil; Drug: Leucovorin; Drug: Irinotecan; Drug: Bevacizumab
- ARM F- BBI608 in combination with Regorafenib (Experimental): BBI608 is administered orally twice daily, continuously. Regorafenib 120 mg will be administered orally once daily, with a low-fat meal and be continued for 21 consecutive days of every 28 days thereafter. If regorafenib is tolerated in the first cycle, dosage may be increased to 160 mg once daily as tolerated after the first cycle.
  Interventions: Drug: BBI608; Drug: Regorafenib
- Arm G- BBI608 in combination with Irinotecan (Experimental): BBI608 is administered orally twice daily, continuously. Irinotecan 180 mg/m^2 will be administered intravenously. This regimen will be repeated every 14 days thereafter.
  Interventions: Drug: BBI608; Drug: Irinotecan

INTERVENTIONS:
Drug: BBI608
  Other Names: Napabucasin; BB608; BBI-608
Drug: Fluorouracil
  Other Names: 5-FU; Carac; Efudex; Fluoroplex; Adrucil
  Arms: ARM A- BBI608 in combination with FOLFOX6; ARM B- BBI608 in combination with FOLFOX6 and Bevacizumab; ARM D- BBI608 in combination with FOLFIRI; ARM E- BBI608 in combination with FOLFIRI and Bevacizumab
Drug: Oxaliplatin
  Other Names: Eloxatin
  Arms: ARM A- BBI608 in combination with FOLFOX6; ARM B- BBI608 in combination with FOLFOX6 and Bevacizumab; ARM C- BBI608 in combination with CAPOX
Drug: Leucovorin
  Other Names: Folinic Acid
  Arms: ARM A- BBI608 in combination with FOLFOX6; ARM B- BBI608 in combination with FOLFOX6 and Bevacizumab; ARM D- BBI608 in combination with FOLFIRI; ARM E- BBI608 in combination with FOLFIRI and Bevacizumab
Drug: Irinotecan
  Other Names: Camptosar
  Arms: ARM D- BBI608 in combination with FOLFIRI; ARM E- BBI608 in combination with FOLFIRI and Bevacizumab; Arm G- BBI608 in combination with Irinotecan
Drug: Bevacizumab
  Other Names: Avastin
  Arms: ARM B- BBI608 in combination with FOLFOX6 and Bevacizumab; ARM E- BBI608 in combination with FOLFIRI and Bevacizumab
Drug: Capecitabine
  Other Names: Xeloda
  Arms: ARM C- BBI608 in combination with CAPOX
Drug: Regorafenib
  Other Names: Stivarga
  Arms: ARM F- BBI608 in combination with Regorafenib

SUMMARY:
This is an open label, multi-center, Phase 1/2 dose escalation study of BBI608 administered in combination with either FOLFOX6 with and without bevacizumab, or CAPOX, or FOLFIRI with and without bevacizumab, or regorafenib, or irinotecan.

DETAILED DESCRIPTION:
This is an open label, multi-center, Phase 1/2 dose escalation study of BBI608 administered in combination with either FOLFOX6 with and without bevacizumab, or CAPOX, or FOLFIRI with and without bevacizumab, or regorafenib, or irinotecan. A study cycle will consist of daily and continuous oral administration of BBI608 for four weeks (28 days) in combination with FOLFOX6 with and without bevacizumab, or CAPOX, or FOLFIRI with and without bevacizumab, or regorafenib, or irinotecan.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. A histologically confirmed solid tumor of the gastrointestinal tract including

   1. Advanced unresectable, metastatic or recurrent colorectal carcinoma (CRC) for which treatment with FOLFOX6 with or without bevacizumab, FOLFIRI with or without bevacizumab, CAPOX, or regorafenib would be acceptable as determined by the Investigator. FOLFIRI/XELIRI-refractory patients with CRC enrolling on the FOLFIRI study arm must have failed treatment with one FOLFIRI pr XELIRI with or without bevacizumab regimen for unresectable or metastatic disease. Treatment failure is defined as progression of disease (clinical or radiologic) during treatment with FOLFIRI with or without bevacizumab or < 3 months after the last dose of treatment with FOLFIRI with or without bevacizumab. Patients with CRC enrolling on the regorafenib arm of this study will have previously received at least two previous lines of therapy for advanced colorectal cancer, and will have previously received treatment with a fluoropyrimidine, oxaliplatin, and irinotecan. Patients with K-ras wild type tumors enrolling on the regorafenib arm will also have previously received either cetuximab or panitumumab.
   2. Hepatocellular carcinoma for which treatment with FOLFOX6 or CAPOX would be acceptable as determined by the Investigator.
   3. Pancreatic adenocarcinoma for which treatment with FOLFOX6, CAPOX, FOLFIRI, or irinotecan would be acceptable as determined by the Investigator.
   4. Cholangiocarcinoma for which treatment with FOLFOX6 or CAPOX would be acceptable as determined by the Investigator.
   5. Gastric, GEJ or esophageal adenocarcinoma for which treatment with FOLFOX6, CAPOX, FOLFIRI, or irinotecan would be acceptable as determined by the Investigator.
3. Patients may be treatment naïve, or may have received standard chemotherapy; including regimens containing a fluoropyrimidine, or oxaliplatin, or irinotecan, or regorafenib, or bevacizumab.
4. ≥18 years of age.
5. Karnofsky performance status score ≥70%.
6. Male or female patients of child-producing potential agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last BBI608 dose.
7. Females of childbearing potential have a negative serum pregnancy test.
8. AST level ≤2.5 x ULN and ALT ≤ 2.5 × ULN. For patients with liver metastases, AST ≤3.5 x ULN, and AST ≤3.5 x ULN may be enrolled if agreed upon by the investigator and medical monitor for the sponsor.
9. Hemoglobin ≥10 g/dl.
10. Total bilirubin level ≤1.5 × ULN.
11. Creatinine ≤1.5 x ULN or creatinine clearance >60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (as determined by Cockcroft-Gault equation).
12. Absolute neutrophil count ≥ 1.5 x 10^9/L.
13. Platelets ≥100 x 10^9/L.
14. Life expectancy estimated at ≥3 months.

Exclusion Criteria:

1. Anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within 7 days of the first dose of BBI608.
2. Major surgery within 4 weeks prior to first dose.
3. Any known untreated brain metastases. Treated subjects must be stable for 4 weeks after completion of that treatment, with image documentation required. Patients must have no clinical symptoms from brain metastases and must be either off steroids or on a stable dose of steroids for at least 2 weeks prior to protocol enrollment. Patients with known leptomeningeal metastases are excluded, even if treated.
4. Pregnant or breastfeeding.
5. Significant gastrointestinal disorder(s) that would, in the opinion of the Principal Investigator, prevent absorption of an orally available agent
6. Unable or unwilling to swallow BBI608 capsules daily.
7. Prior treatment with BBI608.
8. Uncontrolled intercurrent illness
9. For patients to be treated with a regimen containing 5-fluorouracil/leucovorin:

   1. Known hypersensitivity to 5-fluorouracil/leucovorin
   2. Known dihydropyrimidine dehydrogenase (DPD) deficiency
10. For patients to be treated with a regimen containing capecitabine:

    1. Known hypersensitivity to capecitabine
    2. Known dihydropyrimidine dehydrogenase (DPD) deficiency
    3. Significant gastrointestinal disorder(s) that would, in the opinion of the Principal Investigator, prevent absorption of an orally available agent
11. For patients to be treated with a regimen containing oxaliplatin:

    1. Neurosensory neuropathy ≥ grade 2 at baseline
    2. Known hypersensitivity to oxaliplatin or other platinum containing compounds
12. For patients to be treated with a regimen containing irinotecan:

    1. Known hypersensitivity to irinotecan
    2. Abnormal glucuronidation of bilirubin
13. For patients to be treated with a regimen containing bevacizumab:

    1. Current uncontrolled hypertension as well as prior history of hypertensive crisis or hypertensive encephalopathy
    2. History of cardiac disease: congestive heart failure (CHF) > NYHA Class II; active coronary artery disease, myocardial infarction within 6 months prior to study entry; unevaluated new onset angina within 3 months or unstable angina or cardiac arrhythmias requiring anti-arrhythmic therapy
    3. History of arterial thrombotic or embolic events (within 6 months prior to study entry)
    4. Significant vascular disease
    5. Evidence of bleeding diathesis or clinically significant coagulopathy
    6. Major surgical procedure within 28 days, or anticipation of the need for major surgical procedure during the course of the study as well as minor surgical procedure within 7 days prior to study enrollment
    7. Proteinuria at screening as demonstrated by urinalysis with proteinuria ≥ 2+.
    8. History of abdominal fistula, gastrointestinal perforation, peptic ulcer, or intra-abdominal abscess within 6 months
    9. Ongoing serious, non-healing wound, ulcer, or bone fracture
    10. Known hypersensitivity to any component of bevacizumab
    11. History of reversible posterior leukoencephalopathy syndrome (RPLS)
14. For patients to be treated with a regimen containing regorafenib:

    1. History of cardiac disease: congestive heart failure (CHF) > NYHA Class II; active coronary artery disease, myocardial infarction within 6 months prior to study entry; unevaluated new onset angina within 3 months or unstable angina or cardiac arrhythmias requiring anti-arrhythmic therapy
    2. Current uncontrolled hypertension
    3. Interstitial lung disease with ongoing signs and symptoms at the time of screening
    4. History of HIV infection or chronic hepatitis B or C
    5. Active clinically serious infections
    6. History of arterial or embolic events (within 6 months prior to study entry)
    7. Liver cirrhosis ≥ Child-Pugh class B with uncontrolled ascites
    8. History of RPLS
    9. Ongoing serious, non-healing wound, ulcer, or bone fracture
    10. Evidence of bleeding diathesis or a clinically significant coagulopathy
    11. Renal failure requiring hemo- or peritoneal dialysis
    12. Persistent proteinuria of CTCAE grade 3 (>3.5g/24 hours)
    13. Significant gastrointestinal disorder(s) that would, in the opinion of the Principal Investigator, prevent absorption of an orally available agent
    14. Known hypersensitivity to regorafenib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2014-01; Primary Completion 2019-03 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boston Biomedical, Study Director — Sumitomo Pharma America, Inc.
Locations (15):
- United States (14):
  - Mayo Clinic Campus in Arizona, Phoenix, Arizona
  - Florida Cancer Specialists, Fort Myers, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Parkview Research Center, Fort Wayne, Indiana
  - Indiana University Health Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Indiana University Health Arnett Hospital, Lafayette, Indiana
  - Indiana University Health Ball Memorial Hospital, Muncie, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Institute for Translational Oncology Research, Greenville Health System, Greenville, South Carolina
  - Tennessee Oncology - Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology - Nashville, Nashville, Tennessee
- Ottawa Hospital Cancer Center, Ottawa, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 495 participants were enrolled between March 2014 and September 2017.
Pre-assignment Details: Participants who died, withdrew consent to survival follow up or were lost to follow up were considered to have completed the study.
Groups:
- Napabucasin Plus FOLFOX6: All participants who were enrolled to Arm A to receive napabucasin administered orally, twice daily, in combination with FOLFOX6 regimen administered every 14 days. The regimen consisted of oxaliplatin 85 mg/m2 together with leucovorin 400 mg/m2 administered intravenously starting on Day 1 of Cycle 1, after the first daily dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following oxaliplatin/leucovorin infusion, followed by 5-FU 1200 mg/m2/day (total 2400 mg/m2 over 46-48 hours) by continuous intravenous (IV) infusion.
- Napabucasin Plus FOLFOX6 Plus Bevacizumab: All participants who were enrolled to Arm B to receive napabucasin administered orally, twice daily, in combination with FOLFOX6 plus bevacizumab regimen administered every 14 days. The regimen consisted of oxaliplatin 85 mg/m2 together with leucovorin 400 mg/m2 administered intravenously over 2 hours starting on Day1 of Cycle 1, following the first daily dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following oxaliplatin/leucovorin infusion, followed by 5-FU 1200 mg/m2/day (total 2400 mg/m2 over 46-48 hours) by continuous IV infusion. Bevacizumab 5 mg/kg was administered intravenously following the oxaliplatin/leucovorin infusion.
- Napabucasin Plus CAPOX: All participants who were enrolled to Arm C to receive napabucasin administered orally, twice daily, in combination with CAPOX regimen. The CAPOX regimen was administered orally (capecitabine) and by IV (oxaliplatin). Starting on Day 1 of Cycle 1, capecitabine 850 mg/m2 was administered orally BID following the first daily dose of napabucasin for 14 consecutive days and repeated every 21 days. Oxaliplatin 130 mg/m2 was administered intravenously over 2 hours, following the first daily dose of napabucasin starting on Day 1 of Cycle 1 and repeated every 21 days thereafter. If capecitabine was tolerated at the 850 mg/m2 BID dose, the dosage could have been increased to 1000 mg/m2 BID as tolerated after the first cycle.
- Napabucasin Plus FOLFIRI: All participants who were enrolled to Arm D to receive napabucasin administered orally, twice daily, in combination with FOLFIRI regimen. Irinotecan 180 mg/m2 together with leucovorin 400 mg/m2 was administered intravenously starting on Day 1 of Cycle 1, following the first dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5-FU 1200 mg/m2/day (total 2400 mg/m2) by continuous infusion. This regimen was repeated every 14 days thereafter.
- Napabucasin Plus FOLFIRI Plus Bevacizumab: All participants who were enrolled to Arm E to receive napabucasin administered orally, twice daily, in combination with FOLFIRI plus bevacizumab regimen. Irinotecan 180 mg/m2 together with leucovorin 400 mg/m2 was administered intravenously starting on Day 1 of Cycle 1, following the first dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5 FU 1200 mg/m2/day (total 2400 mg/m2) by continuous infusion. Bevacizumab 5 mg/kg was administered intravenously following the irinotecan/leucovorin infusion. This regimen was repeated every 14 days thereafter.
- Napabucasin Plus Regorafenib: All participants who were enrolled to Arm F to receive napabucasin administered orally, twice daily, in combination with regorafenib 120 mg, administered orally once daily with a low-fat meal, starting on Day 1 of Cycle 1 for 21 consecutive days of every 28 days thereafter. If regorafenib was tolerated in the first cycle, the dosage could have been increased to 160 mg once daily as tolerated after the first cycle.
- Napabucasin Plus Irinotecan: All participants who were enrolled to Arm G to receive napabucasin administered orally, twice daily, in combination with irinotecan 180 mg/m2, administered intravenously starting on Day 1 of Cycle 1, following the first dose of napabucasin. This regimen was repeated every 14 days thereafter.
Period: Overall Study
Arm/Group | Napabucasin Plus FOLFOX6 | Napabucasin Plus FOLFOX6 Plus Bevacizumab | Napabucasin Plus CAPOX | Napabucasin Plus FOLFIRI | Napabucasin Plus FOLFIRI Plus Bevacizumab | Napabucasin Plus Regorafenib | Napabucasin Plus Irinotecan
Started | 115 | 41 | 87 | 156 | 40 | 54 | 2
Completed | 115 | 41 | 87 | 156 | 40 | 54 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Napabucasin Plus FOLFOX6 | Napabucasin Plus FOLFOX6 Plus Bevacizumab | Napabucasin Plus CAPOX | Napabucasin Plus FOLFIRI | Napabucasin Plus FOLFIRI Plus Bevacizumab | Napabucasin Plus Regorafenib | Napabucasin Plus Irinotecan | Total
Number analyzed (Participants) | 115 | 41 | 87 | 156 | 40 | 54 | 2 | 495
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.26) | 55.4 (13.54) | 62.7 (11.69) | 58.3 (12.18) | 55.8 (7.25) | 57.5 (11.56) | 73.0 (1.41) | 59.4 (11.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 12 | 32 | 52 | 15 | 28 | 1 | 189
  Male | 66 | 29 | 55 | 104 | 25 | 26 | 1 | 306
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 4 | 3 | 2 | 5 | 0 | 1 | 1 | 16
  Black | 10 | 3 | 8 | 14 | 4 | 4 | 0 | 43
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 99 | 35 | 73 | 134 | 35 | 49 | 1 | 426
  Other | 0 | 0 | 4 | 3 | 1 | 0 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: Assessment of safety of napabucasin administered in combination with either FOLFOX6 with and without bevacizumab, or CAPOX, or FOLFIRI with and without bevacizumab, or regorafenib, or irinotecan in participants with advanced gastrointestinal malignancies by reporting of adverse events and serious adverse events
Time Frame: The time from the date of first treatment, while the patient is taking napabucasin, and for 30 days after stopping therapy, an average of 4 months.
Measure: Count of Participants; unit: Participants
Groups:
- Napabucasin Plus FOLFOX6: Napabucasin administered orally, twice daily, in combination with FOLFOX6 regimen administered every 14 days. The regimen consisted of oxaliplatin 85 mg/m2 together with leucovorin 400 mg/m2 administered intravenously starting on Day 1 of Cycle 1, after the first daily dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following oxaliplatin/leucovorin infusion, followed by 5-FU 1200 mg/m2/day (total 2400 mg/m2 over 46-48 hours) by continuous intravenous (IV) infusion. Patients included in this group received at least one dose of study drug.
- Napabucasin Plus FOLFOX6 Plus Bevacizumab: Napabucasin administered orally, twice daily, in combination with FOLFOX6 plus bevacizumab regimen administered every 14 days. The regimen consisted of oxaliplatin 85 mg/m2 together with leucovorin 400 mg/m2 administered intravenously over 2 hours starting on Day1 of Cycle 1, following the first daily dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following oxaliplatin/leucovorin infusion, followed by 5-FU 1200 mg/m2/day (total 2400 mg/m2 over 46-48 hours) by continuous IV infusion. Bevacizumab 5 mg/kg was administered intravenously following the oxaliplatin/leucovorin infusion. Patients included in this group received at least one dose of study drug.
- Napabucasin Plus CAPOX: Napabucasin administered orally, twice daily, in combination with CAPOX regimen. The CAPOX regimen was administered orally (capecitabine) and by IV (oxaliplatin). Starting on Day 1 of Cycle 1, capecitabine 850 mg/m2 was administered orally BID following the first daily dose of napabucasin for 14 consecutive days and repeated every 21 days. Oxaliplatin 130 mg/m2 was administered intravenously over 2 hours, following the first daily dose of napabucasin starting on Day 1 of Cycle 1 and repeated every 21 days thereafter. If capecitabine was tolerated at the 850 mg/m2 BID dose, the dosage could have been increased to 1000 mg/m2 BID as tolerated after the first cycle. Patients included in this group received at least one dose of study drug.
- Napabucasin Plus FOLFIRI: Napabucasin administered orally, twice daily, in combination with FOLFIRI regimen. Irinotecan 180 mg/m2 together with leucovorin 400 mg/m2 was administered intravenously starting on Day 1 of Cycle 1, following the first dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5-FU 1200 mg/m2/day (total 2400 mg/m2) by continuous infusion. This regimen was repeated every 14 days thereafter. Patients included in this group received at least one dose of study drug.
- Napabucasin Plus FOLFIRI Plus Bevacizumab: Napabucasin administered orally, twice daily, in combination with FOLFIRI plus bevacizumab regimen. Irinotecan 180 mg/m2 together with leucovorin 400 mg/m2 was administered intravenously starting on Day 1 of Cycle 1, following the first dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5 FU 1200 mg/m2/day (total 2400 mg/m2) by continuous infusion. Bevacizumab 5 mg/kg was administered intravenously following the irinotecan/leucovorin infusion. This regimen was repeated every 14 days thereafter. Patients included in this group received at least one dose of study drug.
- Napabucasin Plus Regorafenib: Napabucasin administered orally, twice daily, in combination with regorafenib 120 mg, administered orally once daily with a low-fat meal, starting on Day 1 of Cycle 1 for 21 consecutive days of every 28 days thereafter. If regorafenib was tolerated in the first cycle, the dosage could have been increased to 160 mg once daily as tolerated after the first cycle. Patients included in this group received at least one dose of study drug.
- Napabucasin Plus Irinotecan: Napabucasin administered orally, twice daily, in combination with irinotecan 180 mg/m2, administered intravenously starting on Day 1 of Cycle 1, following the first dose of napabucasin. This regimen was repeated every 14 days thereafter. Patients included in this group received at least one dose of study drug.
Arm/Group | Napabucasin Plus FOLFOX6 | Napabucasin Plus FOLFOX6 Plus Bevacizumab | Napabucasin Plus CAPOX | Napabucasin Plus FOLFIRI | Napabucasin Plus FOLFIRI Plus Bevacizumab | Napabucasin Plus Regorafenib | Napabucasin Plus Irinotecan
Number analyzed (Participants) | 115 | 41 | 87 | 156 | 40 | 54 | 2
Participants | 115 | 41 | 87 | 156 | 40 | 54 | 2

2. Primary Outcome: The Objective Response Rate of Napabucasin Administered in Combination in FOLFIRI in Patients With FOLFIRI/XELIRI-refractory Metastatic Colorectal Cancer
Description: Assessment of the objective response rate (ORR) of napabucasin administered in combination with FOLFIRI in patients with FOLFIRI/XELIRI-refractory metastatic colorectal cancer. The Objective Response Rate (ORR) is the proportion of participants with a complete response or partial response who have measurable disease at baseline imaging.
Time Frame: From the date of first treatment, every 8 weeks, until the date of first documented objective disease progression, up to 24 months
Population: Analysis limited to a subset of group D in which patients had FOLFIRI/XELIRI refractory metastatic colorectal cancer. Patients in this subgroup also had a baseline scan and at least 1 disease assessment following the initiation of therapy.
Measure: Number; unit: percentage of participants
Groups:
- Napabucasin Plus FOLFIRI: Napabucasin administered orally, twice daily, in combination with FOLFIRI regimen. Irinotecan 180 mg/m2 together with leucovorin 400 mg/m2 was administered intravenously starting on Day 1 of Cycle 1, following the first dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5-FU 1200 mg/m2/day (total 2400 mg/m2) by continuous infusion. This regimen was repeated every 14 days thereafter . Patients in this group had a baseline scan and at least one assessment approximately 8 weeks from baseline.
Arm/Group | Napabucasin Plus FOLFIRI
Number analyzed (Participants) | 51
percentage of participants | 0

3. Secondary Outcome: Determination of the Maximum Observed Concentration (Cmax) and Area Under the Plasma Concentration vs. Time Curve (AUClast)
Description: To determine the maximum concentration of napabucasin and the area under the plasma concentration vs. time curve of napabucasin when administered in combination with either FOLFOX6 with and without bevacizumab, or CAPOX, or FOLFIRI with and without bevacizumab, or regorafenib.
Time Frame: Blood samples drawn on days 1, 2, 15, 16, 21, and 22 of the first study cycle
Population: Sponsor's decision to terminate further development of the napabucasin program. Data collection and analysis were therefore not conducted as planned.
Arm/Group | Napabucasin Plus FOLFOX6 | Napabucasin Plus FOLFOX6 Plus Bevacizumab | Napabucasin Plus CAPOX | Napabucasin Plus FOLFIRI | Napabucasin Plus FOLFIRI Plus Bevacizumab | Napabucasin Plus Regorafenib | Napabucasin Plus Irinotecan
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Pharmacodynamics
Description: To determine the response (increase or decrease) of biomarkers from biopsied tumors following the administration of napabucasin
Time Frame: Day 1 of cycle 2
Population: No on-treatment biopsies were performed therefore no pharmacodynamic testing on tumor tissue was conducted.
Arm/Group | Napabucasin Plus FOLFOX6 | Napabucasin Plus FOLFOX6 Plus Bevacizumab | Napabucasin Plus CAPOX | Napabucasin Plus FOLFIRI | Napabucasin Plus FOLFIRI Plus Bevacizumab | Napabucasin Plus Regorafenib | Napabucasin Plus Irinotecan
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Disease Control Rate
Description: To determine the anti-tumor activity (specifically the disease control rate) of napabucasin administered in combination with either FOLFOX6 with and without bevacizumab, or CAPOX, or FOLFIRI with and without bevacizumab, or regorafenib, or irinotecan. Percentage of participants with a documented complete response, partial response and stable disease based on RECIST 1.1.
Time Frame: as for outcome 2
Population: Patients who received at least 1 cycle of study treatment and had at least 1 disease assessment following the initiation of therapy. Patients missing imaging assessment following the initiation of treatment are not included in the assessment for DCR.
Measure: Number; unit: percentage of participants
Groups:
- Napabucasin Plus FOLFOX6: Napabucasin administered orally, twice daily, in combination with FOLFOX6 regimen administered every 14 days. The regimen consisted of oxaliplatin 85 mg/m2 together with leucovorin 400 mg/m2 administered intravenously starting on Day 1 of Cycle 1, after the first daily dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following oxaliplatin/leucovorin infusion, followed by 5-FU 1200 mg/m2/day (total 2400 mg/m2 over 46-48 hours) by continuous intravenous (IV) infusion. Patients in this group had a baseline scan and at least one assessment approximately 8 weeks from baseline.
- Napabucasin Plus FOLFOX6 Plus Bevacizumab: All participants who were enrolled to Arm B to receive napabucasin administered orally, twice daily, in combination with FOLFOX6 plus bevacizumab regimen administered every 14 days. The regimen consisted of oxaliplatin 85 mg/m2 together with leucovorin 400 mg/m2 administered intravenously over 2 hours starting on Day1 of Cycle 1, following the first daily dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following oxaliplatin/leucovorin infusion, followed by 5-FU 1200 mg/m2/day (total 2400 mg/m2 over 46-48 hours) by continuous IV infusion. Bevacizumab 5 mg/kg was administered intravenously following the oxaliplatin/leucovorin infusion. Patients in this group had a baseline scan and at least one assessment approximately 8 weeks from baseline.
- Napabucasin Plus CAPOX: All participants who were enrolled to Arm C to receive napabucasin administered orally, twice daily, in combination with CAPOX regimen. The CAPOX regimen was administered orally (capecitabine) and by IV (oxaliplatin). Starting on Day 1 of Cycle 1, capecitabine 850 mg/m2 was administered orally BID following the first daily dose of napabucasin for 14 consecutive days and repeated every 21 days. Oxaliplatin 130 mg/m2 was administered intravenously over 2 hours, following the first daily dose of napabucasin starting on Day 1 of Cycle 1 and repeated every 21 days thereafter. If capecitabine was tolerated at the 850 mg/m2 BID dose, the dosage could have been increased to 1000 mg/m2 BID as tolerated after the first cycle. Patients in this group had a baseline scan and at least one assessment approximately 8 weeks from baseline.
- Napabucasin Plus FOLFIRI: All participants who were enrolled to Arm D to receive napabucasin administered orally, twice daily, in combination with FOLFIRI regimen. Irinotecan 180 mg/m2 together with leucovorin 400 mg/m2 was administered intravenously starting on Day 1 of Cycle 1, following the first dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5-FU 1200 mg/m2/day (total 2400 mg/m2) by continuous infusion. This regimen was repeated every 14 days thereafter. Patients in this group had a baseline scan and at least one assessment approximately 8 weeks from baseline.
- Napabucasin Plus FOLFIRI Plus Bevacizumab: All participants who were enrolled to Arm E to receive napabucasin administered orally, twice daily, in combination with FOLFIRI plus bevacizumab regimen. Irinotecan 180 mg/m2 together with leucovorin 400 mg/m2 was administered intravenously starting on Day 1 of Cycle 1, following the first dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5 FU 1200 mg/m2/day (total 2400 mg/m2) by continuous infusion. Bevacizumab 5 mg/kg was administered intravenously following the irinotecan/leucovorin infusion. This regimen was repeated every 14 days thereafter. Patients in this group had a baseline scan and at least one assessment approximately 8 weeks from baseline.
- Napabucasin Plus Regorafenib: All participants who were enrolled to Arm F to receive napabucasin administered orally, twice daily, in combination with regorafenib 120 mg, administered orally once daily with a low-fat meal, starting on Day 1 of Cycle 1 for 21 consecutive days of every 28 days thereafter. If regorafenib was tolerated in the first cycle, the dosage could have been increased to 160 mg once daily as tolerated after the first cycle. Patients in this group had a baseline scan and at least one assessment approximately 8 weeks from baseline.
- Napabucasin Plus Irinotecan: All participants who were enrolled to Arm G to receive napabucasin administered orally, twice daily, in combination with irinotecan 180 mg/m2, administered intravenously starting on Day 1 of Cycle 1, following the first dose of napabucasin. This regimen was repeated every 14 days thereafter. Patients in this group had a baseline scan and at least one assessment approximately 8 weeks from baseline.
Arm/Group | Napabucasin Plus FOLFOX6 | Napabucasin Plus FOLFOX6 Plus Bevacizumab | Napabucasin Plus CAPOX | Napabucasin Plus FOLFIRI | Napabucasin Plus FOLFIRI Plus Bevacizumab | Napabucasin Plus Regorafenib | Napabucasin Plus Irinotecan
Number analyzed (Participants) | 75 | 21 | 47 | 105 | 23 | 32 | 1
percentage of participants | 54.7 | 76.2 | 55.3 | 65.7 | 87.0 | 34.4 | 100

6. Secondary Outcome: Disease Control Rate of Patients With FOLFIRI/XELIRI-refractory Metastatic Colorectal Cancer
Description: To determine the disease control rate of napabucasin administered in combination with FOLFIRI in patients with FOLFIRI/XELIRI-refractory metastatic colorectal cancer. Percentage of participants with a documented complete response, partial response and stable disease based on RECIST 1.1.
Time Frame: as for outcome 2
Population: Patients with FOLFIRI/XELIRI refractory metastatic colorectal cancer who received at least 1 cycle of study treatment and had at least 1 disease assessment following the initiation of therapy. Patients missing imaging assessment following the initiation of treatment are not included in the assessment for DCR.
Measure: Number; unit: percentage of participants
Arm/Group | Napabucasin Plus FOLFIRI
Number analyzed (Participants) | 51
percentage of participants | 56.9

7. Secondary Outcome: Progression Free Survival of Patients With FOLFIRI/XELIRI-refractory Metastatic Colorectal Cancer
Description: The effect of napabucasin given in combination with FOLFIRI on Progression Free Survival (PFS) of patients with FOLFIRI/XELIRI-refractory metastatic colorectal cancer. PFS of patients with FOLFIRI/XELIRI-refractory metastatic colorectal cancer.
Time Frame: The time from the date of first treatment to the date of first documentation of disease progression or death due to any cause, up to thirty six months
Population: Analysis limited to a subset of group D in which patients had FOLFIRI/XELIRI refractory metastatic colorectal cancer. Patients in this subgroup also had a baseline scan and at least 1 on study scan or died from any cause.
Measure: Number (95% Confidence Interval); unit: months
Groups:
- Napabucasin Plus FOLFIRI: Napabucasin administered orally, twice daily, in combination with FOLFIRI regimen. Irinotecan 180 mg/m2 together with leucovorin 400 mg/m2 was administered intravenously starting on Day 1 of Cycle 1, following the first dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5-FU 1200 mg/m2/day (total 2400 mg/m2) by continuous infusion. This regimen was repeated every 14 days thereafter. Patients in this group had a baseline scan and at least one on study scan or died from any cause.
Arm/Group | Napabucasin Plus FOLFIRI
Number analyzed (Participants) | 70
months | 20.82 [11.42 to 32.13]

8. Secondary Outcome: Overall Survival of Patients With FOLFIRI/XELIRI-refractory Metastatic Colorectal Cancer
Description: The effect of napabucasin given in combination with FOLFIRI on Overall Survival (OS) of patients with FOLFIRI/XELIRI-refractory metastatic colorectal cancer.
Time Frame: 4 weeks after the patient has been off study treatment, every 3 months thereafter until death, the study closes, up to 36 months.
Population: Analysis limited to a subset of group D in which patients had FOLFIRI/XELIRI refractory metastatic colorectal cancer.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Napabucasin Plus FOLFIRI: Napabucasin administered orally, twice daily, in combination with FOLFIRI regimen. Irinotecan 180 mg/m2 together with leucovorin 400 mg/m2 was administered intravenously starting on Day 1 of Cycle 1, following the first dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5-FU 1200 mg/m2/day (total 2400 mg/m2) by continuous infusion. This regimen was repeated every 14 days thereafter . The patients in this subgroup were assessed to have FOLFIRI/XELIRI refractory metastatic colorectal cancer prior to enrollment.
Arm/Group | Napabucasin Plus FOLFIRI
Number analyzed (Participants) | 70
months | 8.97 [6.80 to 11.76]

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events were assessed from the date of first treatment through 30 days of the last administration of study drug, an average of 4 months. All-Cause Mortality was assessed from the date of first treatment until death, up to 36 months.
Groups:
- Napabucasin Plus FOLFOX6: All participants who received at least 1 dose of napabucasin administered orally, twice daily, in combination with FOLFOX6 regimen administered every 14 days. The regimen consisted of oxaliplatin 85 mg/m2 together with leucovorin 400 mg/m2 administered intravenously starting on Day 1 of Cycle 1, after the first daily dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following oxaliplatin/leucovorin infusion, followed by 5-FU 1200 mg/m2/day (total 2400 mg/m2 over 46-48 hours) by continuous intravenous (IV) infusion.
- Napabucasin Plus FOLFOX6 Plus Bevacizumab: All participants who received at least 1 dose of napabucasin administered orally, twice daily, in combination with FOLFOX6 plus bevacizumab regimen administered every 14 days. The regimen consisted of oxaliplatin 85 mg/m2 together with leucovorin 400 mg/m2 administered intravenously over 2 hours starting on Day1 of Cycle 1, following the first daily dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following oxaliplatin/leucovorin infusion, followed by 5-FU 1200 mg/m2/day (total 2400 mg/m2 over 46-48 hours) by continuous IV infusion. Bevacizumab 5 mg/kg was administered intravenously following the oxaliplatin/leucovorin infusion.
- Napabucasin Plus CAPOX: All participants who received at least 1 dose of napabucasin administered orally, twice daily, in combination with CAPOX regimen. The CAPOX regimen was administered orally (capecitabine) and by IV (oxaliplatin). Starting on Day 1 of Cycle 1, capecitabine 850 mg/m2 was administered orally BID following the first daily dose of napabucasin for 14 consecutive days and repeated every 21 days. Oxaliplatin 130 mg/m2 was administered intravenously over 2 hours, following the first daily dose of napabucasin starting on Day 1 of Cycle 1 and repeated every 21 days thereafter. If capecitabine was tolerated at the 850 mg/m2 BID dose, the dosage could have been increased to 1000 mg/m2 BID as tolerated after the first cycle.
- Napabucasin Plus FOLFIRI: All participants who received at least 1 dose of napabucasin administered orally, twice daily, in combination with FOLFIRI regimen. Irinotecan 180 mg/m2 together with leucovorin 400 mg/m2 was administered intravenously starting on Day 1 of Cycle 1, following the first dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5-FU 1200 mg/m2/day (total 2400 mg/m2) by continuous infusion. This regimen was repeated every 14 days thereafter.
- Napabucasin Plus FOLFIRI Plus Bevacizumab: All participants who received at least 1 dose of napabucasin administered orally, twice daily, in combination with FOLFIRI plus bevacizumab regimen. Irinotecan 180 mg/m2 together with leucovorin 400 mg/m2 was administered intravenously starting on Day 1 of Cycle 1, following the first dose of napabucasin. A 5-FU 400 mg/m2 bolus was administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5 FU 1200 mg/m2/day (total 2400 mg/m2) by continuous infusion. Bevacizumab 5 mg/kg was administered intravenously following the irinotecan/leucovorin infusion. This regimen was repeated every 14 days thereafter.
- Napabucasin Plus Regorafenib: All participants who received at least 1 dose of napabucasin administered orally, twice daily, in combination with regorafenib 120 mg, administered orally once daily with a low-fat meal, starting on Day 1 of Cycle 1 for 21 consecutive days of every 28 days thereafter. If regorafenib was tolerated in the first cycle, the dosage could have been increased to 160 mg once daily as tolerated after the first cycle.
- Napabucasin Plus Irinotecan: All participants who received at least 1 dose of napabucasin administered orally, twice daily, in combination with irinotecan 180 mg/m2, administered intravenously starting on Day 1 of Cycle 1, following the first dose of napabucasin. This regimen was repeated every 14 days thereafter.
Arm/Group | Napabucasin Plus FOLFOX6 | Napabucasin Plus FOLFOX6 Plus Bevacizumab | Napabucasin Plus CAPOX | Napabucasin Plus FOLFIRI | Napabucasin Plus FOLFIRI Plus Bevacizumab | Napabucasin Plus Regorafenib | Napabucasin Plus Irinotecan
All-Cause Mortality (participants affected / at risk) | 104/115 | 31/41 | 82/87 | 129/156 | 33/40 | 50/54 | 2/2
Serious Adverse Events (participants affected / at risk) | 52/115 | 10/41 | 40/87 | 58/156 | 16/40 | 23/54 | 2/2
Other Adverse Events (participants affected / at risk) | 115/115 | 41/41 | 87/87 | 156/156 | 40/40 | 54/54 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Napabucasin Plus FOLFOX6 (N=115) | Napabucasin Plus FOLFOX6 Plus Bevacizumab (N=41) | Napabucasin Plus CAPOX (N=87) | Napabucasin Plus FOLFIRI (N=156) | Napabucasin Plus FOLFIRI Plus Bevacizumab (N=40) | Napabucasin Plus Regorafenib (N=54) | Napabucasin Plus Irinotecan (N=2)
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 5 | 0 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 5 | 4 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0 | 9 | 4 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 3 | 5 | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 3 | 1 | 3 | 1 | 6 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Large instestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Megacolon (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 4 | 0 | 1 | 4 | 0 | 1 | 0
Disease progression (General disorders) | 2 | 0 | 5 | 3 | 0 | 2 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage intranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
syncope (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1
migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 1 | 7 | 3 | 2 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 4 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 4 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 5 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 6 | 0 | 5 | 3 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 1 | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 1 | 3 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Salmonella sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyuria (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
pelvic fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0
subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0
gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
embolism (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
pelvic venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0 | 0 | 0 | 0
pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Napabucasin Plus FOLFOX6 (N=115) | Napabucasin Plus FOLFOX6 Plus Bevacizumab (N=41) | Napabucasin Plus CAPOX (N=87) | Napabucasin Plus FOLFIRI (N=156) | Napabucasin Plus FOLFIRI Plus Bevacizumab (N=40) | Napabucasin Plus Regorafenib (N=54) | Napabucasin Plus Irinotecan (N=2)
Diarrhoea (Gastrointestinal disorders) | 94 | 37 | 75 | 139 | 39 | 42 | 1
Nausea (Gastrointestinal disorders) | 87 | 32 | 63 | 100 | 37 | 26 | 2
Vomiting (Gastrointestinal disorders) | 66 | 25 | 49 | 76 | 32 | 16 | 1
Abdominal pain (Gastrointestinal disorders) | 61 | 22 | 37 | 58 | 22 | 26 | 2
Stomatitis (Gastrointestinal disorders) | 12 | 5 | 2 | 12 | 12 | 2 | 0
Constipation (Gastrointestinal disorders) | 27 | 11 | 18 | 31 | 14 | 15 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 3 | 7 | 11 | 5 | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 10 | 2 | 9 | 9 | 6 | 5 | 0
Ascites (Gastrointestinal disorders) | 11 | 3 | 11 | 6 | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 7 | 6 | 2 | 8 | 7 | 3 | 0
Flatulence (Gastrointestinal disorders) | 5 | 2 | 6 | 10 | 6 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 11 | 1 | 2 | 7 | 3 | 4 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 5 | 4 | 5 | 5 | 3 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 3 | 4 | 7 | 5 | 3 | 0
Fatigue (General disorders) | 82 | 25 | 53 | 92 | 33 | 29 | 2
Mucosal inflammation (General disorders) | 15 | 6 | 9 | 11 | 14 | 8 | 0
Pyrexia (General disorders) | 19 | 6 | 13 | 24 | 6 | 10 | 1
Oedema peripheral (General disorders) | 23 | 2 | 12 | 21 | 6 | 3 | 0
Chills (General disorders) | 5 | 7 | 9 | 8 | 3 | 6 | 0
Temperature intolerance (General disorders) | 15 | 4 | 15 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 9 | 3 | 11 | 6 | 2 | 3 | 0
Neuropathy peripheral (Nervous system disorders) | 35 | 13 | 13 | 5 | 6 | 4 | 0
Headache (Nervous system disorders) | 10 | 6 | 9 | 12 | 10 | 7 | 0
Dysgeusia (Nervous system disorders) | 15 | 5 | 13 | 8 | 6 | 4 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 19 | 9 | 14 | 3 | 4 | 1 | 0
Dizziness (Nervous system disorders) | 13 | 5 | 7 | 11 | 2 | 6 | 0
Dehydration (Metabolism and nutrition disorders) | 21 | 10 | 24 | 28 | 6 | 13 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 24 | 8 | 19 | 31 | 9 | 12 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 12 | 2 | 5 | 7 | 2 | 3 | 0
Neutrophil count decreased (Investigations) | 27 | 4 | 3 | 23 | 7 | 2 | 0
Weight decreased (Investigations) | 25 | 10 | 17 | 21 | 13 | 7 | 0
Urine ketone body present (Investigations) | 8 | 7 | 7 | 13 | 8 | 0 | 0
Blood bilirubin increased (Investigations) | 7 | 4 | 6 | 12 | 2 | 7 | 0
Platelet count decreased (Investigations) | 17 | 3 | 4 | 9 | 2 | 2 | 0
Urine leukocyte esterase positive (Investigations) | 6 | 6 | 7 | 10 | 5 | 0 | 0
White blood cell count decreased (Investigations) | 14 | 3 | 2 | 11 | 2 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 8 | 5 | 5 | 4 | 1 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 20 | 15 | 4 | 38 | 14 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 29 | 9 | 15 | 40 | 9 | 10 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 8 | 18 | 19 | 4 | 6 | 0
Lymphopenia (Blood and lymphatic system disorders) | 7 | 5 | 4 | 5 | 4 | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 7 | 5 | 4 | 5 | 4 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 7 | 9 | 16 | 9 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 3 | 3 | 9 | 10 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 4 | 6 | 8 | 0 | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3 | 3 | 6 | 3 | 8 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 8 | 4 | 5 | 4 | 0
Chromaturia (Renal and urinary disorders) | 15 | 3 | 10 | 23 | 7 | 4 | 0
Proteinuria (Renal and urinary disorders) | 6 | 7 | 5 | 15 | 7 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 4 | 3 | 27 | 22 | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 1 | 9 | 3 | 2 | 13 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 2 | 4 | 5 | 6 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 6 | 12 | 29 | 12 | 13 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 8 | 6 | 22 | 10 | 7 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 3 | 8 | 6 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 1 | 3 | 9 | 2 | 0
Urinary tract infection (Infections and infestations) | 14 | 3 | 4 | 20 | 9 | 6 | 0
Insomnia (Psychiatric disorders) | 10 | 5 | 5 | 17 | 12 | 7 | 0
Anxiety (Psychiatric disorders) | 11 | 5 | 3 | 8 | 5 | 4 | 0
Depression (Psychiatric disorders) | 13 | 3 | 5 | 6 | 3 | 3 | 0
Hypertension (Vascular disorders) | 6 | 6 | 2 | 3 | 6 | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT02024607/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT02024607/SAP_001.pdf